CLINICAL TRIAL: NCT06415422
Title: Platelet Activity Monitoring for Patients Under Adp Medication Using Verify Now in Subdural Hematoma
Acronym: PAPAYE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 29BRC22.0226
Record Dates: First submitted 2024-05-03; First posted 2024-05-16 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Hematoma, Subdural
MeSH Terms: conditions — Hematoma, Subdural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Daily Sampling in Platelet Function (Other): The management of patients included in this study is not altered from the standard recommended care. The only exception is the daily blood draw into a dry tube for decentralized analysis using VeriFyNow until the normalization of platelet function, which is not part of routine care.
  Interventions: Biological: Biological samples

INTERVENTIONS:
Biological: Biological samples — Biological samples are taken from the patient's catheter inserted upon admission (the usual access route for patients): A daily sample is collected into a dry tube for off-site analysis by VeriFyNow until platelet function normalizes (for example, if platelet function normalizes on Day 2, no further VeriFyNow analysis will be conducted on subsequent days).

SUMMARY:
The brain is encased in three membranes: the pia mater, arachnoid, and dura mater. A subdural hematoma is often a post-traumatic accumulation of blood between the dura mater and the brain, occurring when a trauma tears a small vein on the brain. As the hematoma expands, it compresses the brain, potentially leading to severe neurological symptoms that may require urgent surgical removal. Patients on antiplatelet therapy are at increased risk of larger subdural hematomas and higher morbidity.

The reversibility of antiplatelet effects and the potential benefits of platelet transfusions to halt hematoma expansion or prevent significant re-bleeding during surgical management are still debated. The French Society of Anesthesia and Intensive Care (SFAR) recommends delaying neurosurgical interventions by 5 days if clinically tolerable, with platelet transfusions provided for urgent surgeries within this period. However, prolonged cessation of antithrombotic treatments increases the risk of perioperative thrombotic events.

Literature also notes individual variability in the effectiveness of antiplatelet treatments. European guidelines suggest using platelet function analysis devices alongside standard laboratory coagulation monitoring in trauma patients suspected of platelet dysfunction (Level 2C). The 2019 SFAR guidelines for the emergency management of patients on antiplatelets do not recommend these devices outside of cardiovascular surgery due to a lack of studies.

DETAILED DESCRIPTION:
The brain is encased in three membranes: the pia mater, arachnoid, and dura mater. A subdural hematoma is often a post-traumatic accumulation of blood between the dura mater and the brain, occurring when a trauma tears a small vein on the brain. As the hematoma expands, it compresses the brain, potentially leading to severe neurological symptoms that may require urgent surgical removal. Patients on antiplatelet therapy are at increased risk of larger subdural hematomas and higher morbidity.

The reversibility of antiplatelet effects and the potential benefits of platelet transfusions to halt hematoma expansion or prevent significant re-bleeding during surgical management are still debated. The French Society of Anesthesia and Intensive Care (SFAR) recommends delaying neurosurgical interventions by 5 days if clinically tolerable, with platelet transfusions provided for urgent surgeries within this period. However, prolonged cessation of antithrombotic treatments increases the risk of perioperative thrombotic events.

Literature also notes individual variability in the effectiveness of antiplatelet treatments. European guidelines suggest using platelet function analysis devices alongside standard laboratory coagulation monitoring in trauma patients suspected of platelet dysfunction (Level 2C). The 2019 SFAR guidelines for the emergency management of patients on antiplatelets do not recommend these devices outside of cardiovascular surgery due to a lack of studies.

ELIGIBILITY:
Inclusion Criteria:

Patient >18 years old Patient managed for a subdural hematoma in neurosurgery or intensive care under Acetylsalicylic Acid (aspirin) regardless of the dose.

No objection from the patient

Exclusion Criteria:

Patient under effective anticoagulation or on antiplatelet therapy other than acetylsalicylic acid (combination of two antiplatelets) Pregnant or breastfeeding woman Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Platelet Function Progression | Day 0
  Evaluation of the difference between the time to achieve functional platelets, measured by the analysis of platelet function and the recommended management delay by SFAR of 5 days after the cessation of the antiplatelet drug
Evaluation of Platelet Function Progression | Day 1
  Evaluation of the difference between the time to achieve functional platelets, measured by the analysis of platelet function and the recommended management delay by SFAR of 5 days after the cessation of the antiplatelet drug
Evaluation of Platelet Function Progression | Day 2
  Evaluation of the difference between the time to achieve functional platelets, measured by the analysis of platelet function and the recommended management delay by SFAR of 5 days after the cessation of the antiplatelet drug
Evaluation of Platelet Function Progression | Day 3
  Evaluation of the difference between the time to achieve functional platelets, measured by the analysis of platelet function (defined by the time elapsed between the last intake of antiplatelet drugs and the normalization of platelet function measured by VeriFyNow), and the recommended management delay by SFAR of 5 days after the cessation of the antiplatelet drug
  An analysis of the kinetics of recovery of platelet function in patients on aspirin managed for a subdural hematoma will be conducted to assess this criterion.
Evaluation of Platelet Function Progression | Day 4
  Evaluation of the difference between the time to achieve functional platelets, measured by the analysis of platelet function and the recommended management delay by SFAR of 5 days after the cessation of the antiplatelet drug
Evaluation of Platelet Function Progression | Day 5
  Evaluation of the difference between the time to achieve functional platelets, measured by the analysis of platelet function and the recommended management delay by SFAR of 5 days after the cessation of the antiplatelet drug

SECONDARY OUTCOMES:
Comparison of platelet function measurement between calculation and VerifyNow | Day 0
  Comparison of platelet function measurement calculated by the theoretical formula based on the patient's initial platelet count and a 10% daily platelet turnover rate, and the VeriFyNow.
Comparison of platelet function measurement between calculation and VerifyNow | Day 1
  Comparison of platelet function measurement calculated by the theoretical formula based on the patient's initial platelet count and a 10% daily platelet turnover rate, and the VeriFyNow.
Comparison of platelet function measurement between calculation and VerifyNow | Day 2
  Comparison of platelet function measurement calculated by the theoretical formula based on the patient's initial platelet count and a 10% daily platelet turnover rate, and the VeriFyNow.
Comparison of platelet function measurement between calculation and VerifyNow | Day 3
  Comparison of platelet function measurement calculated by the theoretical formula based on the patient's initial platelet count and a 10% daily platelet turnover rate, and the VeriFyNow.
Comparison of platelet function measurement between calculation and VerifyNow | Day 4
  Comparison of platelet function measurement calculated by the theoretical formula based on the patient's initial platelet count and a 10% daily platelet turnover rate, and the VeriFyNow.
Comparison of platelet function measurement between calculation and VerifyNow | Day 5
  Comparison of platelet function measurement calculated by the theoretical formula based on the patient's initial platelet count and a 10% daily platelet turnover rate, and the VeriFyNow.
Comparison of the actual surgical management time with the theoretical formula-based time | Immediately after intervention
  Description and comparison of the actual surgical management time and the time to achieve functional platelets calculated by the theoretical formula based on the initial platelet count of the patient and a 10% daily platelet turnover rate.
Evaluation of Incidence of Platelet Transfusion | Day 0
  Evaluation of the Incidence of Platelet Transfusion on Actual Surgical Management Time
Evaluation of Incidence of Platelet Transfusion | Day 1
  Evaluation of the Incidence of Platelet Transfusion on Actual Surgical Management Time
Evaluation of Incidence of Platelet Transfusion | Day 2
  Evaluation of the Incidence of Platelet Transfusion on Actual Surgical Management Time
Evaluation of Incidence of Platelet Transfusion | Day 3
  Evaluation of the Incidence of Platelet Transfusion on Actual Surgical Management Time
Evaluation of Incidence of Platelet Transfusion | Day 4
  Evaluation of the Incidence of Platelet Transfusion on Actual Surgical Management Time
Evaluation of Incidence of Platelet Transfusion | Day 5
  Evaluation of the Incidence of Platelet Transfusion on Actual Surgical Management Time
Comparison of the total duration of antiplatelet cessation | Day 0
  Comparison of the total duration of antiplatelet cessation (from preoperative stop to resumption validated by neurosurgeons) between actual management and optimal management.
Comparison of the total duration of antiplatelet cessation | Day 1
  Comparison of the total duration of antiplatelet cessation (from preoperative stop to resumption validated by neurosurgeons) between actual management and optimal management.
Comparison of the total duration of antiplatelet cessation | Day 2
  Comparison of the total duration of antiplatelet cessation (from preoperative stop to resumption validated by neurosurgeons) between actual management and optimal management.
Comparison of the total duration of antiplatelet cessation | Day 3
  Comparison of the total duration of antiplatelet cessation (from preoperative stop to resumption validated by neurosurgeons) between actual management and optimal management.
Comparison of the total duration of antiplatelet cessation | Day 4
  Comparison of the total duration of antiplatelet cessation (from preoperative stop to resumption validated by neurosurgeons) between actual management and optimal management.
Comparison of the total duration of antiplatelet cessation | Day 5
  Comparison of the total duration of antiplatelet cessation (from preoperative stop to resumption validated by neurosurgeons) between actual management and optimal management.
Evaluation of cardiovascular complications | Month 3
  Evaluation of the number of cardiovascular complications occurring within 6 months (acute coronary syndrome, ischemic stroke, thrombophlebitis, or pulmonary embolism)
Evaluation of cardiovascular complications | Month 6
  Evaluation of the number of cardiovascular complications occurring within 6 months (acute coronary syndrome, ischemic stroke, thrombophlebitis, or pulmonary embolism)
Evaluation of the mRs score | Immediately after discharge
  Evaluation of the mRs (modified Rankin Scale) score at discharge from the neurosurgery department, and at 3 and 6 months.
Evaluation of the mRs score | Month 3
  Evaluation of the mRs (modified Rankin Scale) score at discharge from the neurosurgery department, and at 3 and 6 months.
Evaluation of the mRs score | Month 6
  Evaluation of the mRs (modified Rankin Scale) score at discharge from the neurosurgery department, and at 3 and 6 months.

IPD SHARING:
Plan to Share IPD: Undecided